CLINICAL TRIAL: NCT06105073
Title: "Effect of a Pulmonary Rehabilitation Program in Patients With Interstitial Lung Disease Associated With Systemic Sclerosis on Oxygen Consumption, Functionality, and Quality of Life"
Brief Title: "Pulmonary Rehabilitation Program in Patients With Interstitial Lung Disease Associated With Systemic Sclerosis"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Other Study IDs: CNCI-R-2021-785-064
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-10

CONDITIONS: Systemic Sclerosis Associated Interstitial Lung Disease
Keywords: Systemic sclerosis; Interstitial lung disease; Pulmonary rehabilitation program; Quality of life; Oxygen consumption; Functionality
MeSH Terms: conditions — Scleroderma, Systemic; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients whit Systemic Sclerosis asociated Interstitial Lung Disease: Consecutive patients who attend the Rheumatology and Internal Medicine services with a confirmed diagnosis of Systemic Sclerosis associated Interstitial Lung disease, from the Medical Center, La Raza IMSS.
  Interventions: Procedure: Pulmonary Rehabilitation Program

INTERVENTIONS:
Procedure: Pulmonary Rehabilitation Program — Consecutive patients who attend with a confirmed diagnosis of Systemic Sclerosis associated Interstitial Lung disease, at the Speciality Hospital from the Medical Center La Raza IMSS. The anxiety and depression questionnaire will be applied to them. Goldberg, as well as the SF-36 questionnaire to evaluate quality of life and the SySQ questionnaire to evaluate functionality, to include these data in the analysis, these questionnaires are validated in our population and have been widely used. All participants (T0) will undergo Forced Spirometry, Carbon Monoxide Diffusion Capacity and Cardiopulmonary Exercise Test. Then they will enter a supervised pulmonary rehabilitation program that consists of 36 sessions, which is equivalent to 12 weeks. At the end of this period (T1), again the respiratory function tests (spirometry, DLCO and Cardiopulmonary Exercise Test) as well as the Goldberg, SF-36 and SySq questionnaires.

SUMMARY:
Interstitial Lung Disease associated with Systemic Sclerosis currently represents the main cause of death in this disease, it is also the cause of significant morbidity, which is why pulmonary rehabilitation strategies can be of great benefit in this group of patients. The aim of this study is to determine the effect of a 36-session supervised pulmonary rehabilitation program compared before and after, on oxygen consumption, functionality, and quality of life in Interstitial Lung

The main question it aims to answer are:

What effect will have with a 36-session supervised pulmonary rehabilitation program, compared before and after, on oxygen consumption, functionality and quality of life in Interstitial Lung Disease associated with Systemic Sclerosis, estimated by Cardiopulmonary Exercise Test, the questionnaire self-administered SySQ (systemic sclerosis functionality questionnaire) and the self-administered questionnaire SF-36.

Disease associated with Systemic Sclerosis. Study design: Quasi-experimental, longitudinal, comparative before and after study. Methods: Consecutive patients who attend the Rheumatology and Internal Medicine services with a confirmed diagnosis of Systemic Sclerosis, at the Speciality Hospital of the National Medical Center La raza IMSS (Mexican Institute of Social Security), all those patients who wish to participate in the study will be asked to sign the informed consent letter, subsequently the Goldberg anxiety and depression questionnaire will be applied, as well as the SF-36 questionnaire to evaluate quality of life and SySQ to evaluate functionality, all participants will undergo Forced Spirometry, Carbon Monoxide Diffusion Capacity and Cardiopulmonary Exercise Test, the Pulmonary Function laboratory of the General Hospital National Medical Center La Raza IMSS . Subsequently, they will be sent to the Pulmonary Rehabilitation service, where they will enter a supervised pulmonary rehabilitation program that consists of 36 sessions (12 weeks). After the end of the program, respiratory function tests and tests will be performed again questionnaires, pulmonary function tests and cardiopulmonary exercise test.

DETAILED DESCRIPTION:
Consecutive patients who attend the Rheumatology and Internal Medicine services with a confirmed diagnosis of Interstitial Lung Disease associated Systemic Sclerosis, at the Speciality Hospital from the National Medical Center La Raza IMSS, all patients who wish to participate in the study will be asked to sign the informed consent letter from the participating researchers, subsequently the anxiety and depression questionnaire will be applied to them. Goldberg, as well as the SF-36 questionnaire to evaluate quality of life and the SySQ questionnaire to evaluate functionality, to include these data in the analysis, as well as history of smoking, occupational and environmental exposures to both biomass combustion smoke and inorganic powders, these questionnaires are validated in our population and have been widely used, the data corresponding to the time of evolution of the disease, medications used, comorbidities and levels of antibodies and acute phase reactants will be collected from the clinical records. of each of the participants. All participants (T0) will undergo Forced Spirometry, Carbon Monoxide Diffusion Capacity (DLCO) and Cardiopulmonary Exercise Test. The Pulmonary Function Laboratory of the National Medical Center General Hospital has qualified and trained personnel in performing respiratory function tests, the interpretation of said results will be carried out by the main author (doctoral student) who has a high specialty in Respiratory Physiology and Pulmonary Function Laboratory. Subsequently, the patients will be sent to the Pulmonary Rehabilitation service of the La Raza National Medical Center where they will enter a supervised pulmonary rehabilitation program that consists of 36 sessions, which is equivalent to 12 weeks. At the end of this period (T1), again the respiratory function tests (spirometry, plethysmography, DLCO, arterial blood gases and Cardiopulmonary Exercise Test) as well as the Goldberg, SF-36 and SySq questionnaires. The protocol has been submitted for approval to the National Health Research Committee (CNCI).

Study procedures. Every day prior to the start of the work day in the Pulmonary Function Laboratory of the National Medical Center La Raza IMSS, the cleaning and disinfection procedures of the equipment are carried out according to the manufacturer's requirements and the procedures are carried out. calibration, both for volume and flow linearity according to ATS/ERS 2005 standards for flow sensors, as well as linearity calibrations for the gas analyzer and pressure and temperature calibrations of the equipment.

Prior to performing the lung function tests, anthropometric measurements will be performed as follows:

* Height: with the patient in a standing position, height will be obtained with a wall stadiometer model 206 (Seca GMBH & Co., Hamburg, Germany). This measurement will be carried out by placing the heels together, close to the wall, as well as the calves, buttocks, shoulder blades and head. The head will be positioned by asking the patient to look forward, keeping the lateral canthus of the orbit horizontal in relation to the auditory meatus (Frankfort plane).
* Weight: with the patient wearing light clothing, the weight will be obtained using a precision digital scale model 813 (Seca GMBH & Co., Hamburg, Germany).

Goldberg Questionnaire for Anxiety and Depression The Goldberg Anxiety and Depression Scale is both a screening test, with healthcare and epidemiological uses, and an interview guide. It is a test that not only guides the diagnosis towards anxiety or depression (or both in mixed cases), but also discriminates between them and measures their respective intensities.

The Goldberg Anxiety and Depression Scale contains 2 subscales with nine questions in each: anxiety subscale (questions 1-9) and depression subscale (questions 10-18). The first 4 questions of each subscale (questions 1-4) and (questions 10-13), respectively, act as a precondition to determine whether the rest of the questions should be attempted. Specifically, if a minimum of 2 questions from questions 1-4 are not answered affirmatively, the rest of the questions in the first subscale should not be answered, while in the case of the second subscale it is sufficient to answer affirmatively to one question. between questions 10-13 to be able to proceed to answer the rest of the questions.

The cut-off points are 4 or more for the anxiety subscale and 2 or more for the depression subscale, with scores being higher the more serious the problem is (the maximum possible being 9 in each of the subscales). Even when the questions are very clear, the answers only admit dichotomy, so that sometimes, when coincidences of slight intensity are involved, the judgment of a specialist professional is necessary to assess the clinical significance of the answer.

SF-36 Questionnaire This questionnaire contains 36 items to measure health in eight dimensions: perception of general health, physical and social functioning, limitations of function due to physical or emotional problems, health, vitality and body pain. For each dimension, items are coded, summed, and transformed into a scale from 0 (worst health) to 100 (best health). The eight dimensions can be reduced to two summary measures, a physical component score (PCS) and a mental component score (MCS). The MCID in brief form 36 (SF-36) has been estimated in patients with rheumatoid arthritis which has been estimated at 20% improvement in baseline score.

SySQ Questionnaire. It is a self-administered functionality questionnaire for SSc (Systemic Sclerosis Questionnaire [SySQ]), which assesses the difficulty in carrying out activities of daily living and the intensity and frequency of the symptoms with the greatest functional impact in SSc. This instrument was originally designed in German and has been validated in Spanish by this working group. Include 3 domains concerning activities of daily living, intensity and frequency of symptoms. Three domains in 4 categories: 1) general symptoms; 2) musculoskeletal symptoms; 3) cardiopulmonary symptoms, and 4) symptoms of the digestive tract, which are the main organs affected and represent the greatest impact on the functionality of patients with Ssc. This scale includes an ability to perform an action section (0 = no difficulty, 1 = some difficulty, 2 = some difficulty, 3 = unable to do); another section describes the intensity of the symptoms (0 = no, 1 = mild, 2 = moderate, 3 = very severe), and finally there is a section on the frequency of the symptoms (0 = no, 1 = sometimes, 2 = often, 3 = always). The final score of the scale is calculated by averaging the maximum value obtained in each domain (block of questions) divided by 3 (given that there are 3 domains), and that value goes from 0 (normal functionality) to 3 (minimal functionality). The questionnaire formats will be provided by the pulmonary function laboratory staff to the study participants.

Forced spirometry. Spirometry is the main test of respiratory function, it evaluates respiratory mechanics and is the standard for diagnosing bronchial obstruction. The test was performed in accordance with ATS/ERS 2005 standards. Once the patient is prepared for the test, the patient is instructed about the procedure. It is explained to him that he will be sitting (preferably in a fixed chair with arm support), with his trunk upright and his head slightly elevated; He is instructed to place a mouthpiece and a nose clip in his mouth and to perform a maximum inhalation and then an exhalation with an explosive and sustained onset. The maneuver will be carried out in a closed circuit. The patient will be asked to maintain forced expiration for at least 6 seconds until reaching a plateau of at least 1 second. The available equipment is the brand and model Jaeger Sentry Suite Ver. 2.13, IOS, Germany.

Carbon monoxide diffusing capacity (DLCO) This test is necessary to evaluate gas transfer, it is necessary to complement the diagnosis and rule out interstitial damage in patients who present restriction of extrapulmonary origin. The test will be performed according to ATS/ERS 2017 standards. The patient will be seated (fixed chair with arm support), with the trunk upright and the head slightly elevated. You will be fitted with a nose clip and asked to breathe into the equipment through a sterile antibacterial mouthpiece. At the beginning, breaths were performed in tidal volume and later, based on residual functional capacity, a maximum expiration was made, until reaching a plateau of 1 second and reaching residual volume. When the residual volume was reached, the valves were activated. The patient was encouraged to perform maximum and rapid inspiration (less than 3 seconds), which reached more than 90% of his vital capacity. He must maintain an apnea for 10 seconds, taking care that there are no leaks or valsalva maneuver. The patient was instructed to make a maximum expiration, but slowly and relaxed, lasting longer than 4 seconds. The time between maneuvers was at least 4 minutes. A minimum of two efforts were completed with acceptability criteria in accordance with ATS/ERS 2017. The available equipment is the brand and model Jaeger Sentry Suite Ver. 2.13, Germany. Exercise test.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of SSc, determined by the treating rheumatology service either from the Rheumatology and/or Internal Medicine Service of the Specialty Hospital of the National Medical Center La Raza IMSS , based on the ACR/EULAR 2013 criteria for SSc.
* Time of evolution of the disease indistinct. You can be treated with any of the drugs in the spectrum of autoimmune disease treatment (immunosuppressants, steroids, biologics, etc.).
* Diagnosis of Interstitial Lung Disease associated with SSc, confirmed by HRCT and FVC < 80% or TLC < 80% or DLCO < 80%.

Exclusion Criteria:

* Pregnant
* Chest, abdominal pain, oral or facial pain that prevents using the mouthpiece or forced expiration.
* Stress incontinence, dementia or confusion.
* Who have contraindications for performing physical effort.
* Oxygen dependence that does not allow its withdrawal for more than 10 minutes.
* Recent surgeries less than 1 month in case of thorax and upper abdomen and less than three months in case of retina and middle ear surgery.
* Belonging to vulnerable groups (homeless people, prisoners, etc.)
* Failure to obtain the informed consent signature
* Presence of contraindication to exercise such as muscular or orthopedic injuries.
* Who have presented disease activity data that would have required a change in pharmacological treatment in a period of less than 12 weeks prior to the start of the rehabilitation program.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who come to the Rheumatology and Internal Medicine services with a confirmed diagnosis of Interstitial Lung Disease associated Systemic Sclerosis from the National Medical Center La Raza IMSS
Sampling Method: Non-Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Oxygen consumption peak | It will be measured before the pulmonary rehabilitation therapy and at the end (12 weeks), estimated by cardiopulmonary exercise test
  Change in oxygen consumption of at least 1.15 ml/kg/min relative to the measurement before receiving the supervised pulmonary rehabilitation program, measured in ml/min.
Quality of life health related | It will be measured before the pulmonary rehabilitation therapy and at the end (12 weeks)
  Change in the score obtained in the SF36 quality of life questionnaire of at least 20% in relation to the baseline score obtained before receiving the 12-week supervised pulmonary rehabilitation program. Where 0 is the worst quality of life and 100 is the best quality of life, scores below 50 are considered poor quality of life.
Functionality | t will be measured before the pulmonary rehabilitation therapy and at the end (12 weeks)
  Change of 1 category in the score of the functionality scale for systemic sclerosis SySQ, in relation to the score obtained before entering the 12-week supervised pulmonary rehabilitation program.
  This scale includes an ability to perform an action section (0 = no difficulty, 1 = some difficulty, 2 = some difficulty, 3 = unable to do); another section describes the intensity of the symptoms (0 = no, 1 = mild, 2 = moderate, 3 = very severe), and finally there is a section on the frequency of the symptoms (0 = no, 1 = sometimes, 2 = often, 3 = always). The final score of the scale is calculated by averaging the maximum value obtained in each domain (block of questions) divided by 3 (given that there are 3 domains), and that value goes from 0 (normal functionality) to 3 (minimal functionality)

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Medico Nacional La Raza, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van den Hoogen F, Khanna D, Fransen J, Johnson SR, Baron M, Tyndall A, Matucci-Cerinic M, Naden RP, Medsger TA Jr, Carreira PE, Riemekasten G, Clements PJ, Denton CP, Distler O, Allanore Y, Furst DE, Gabrielli A, Mayes MD, van Laar JM, Seibold JR, Czirjak L, Steen VD, Inanc M, Kowal-Bielecka O, Muller-Ladner U, Valentini G, Veale DJ, Vonk MC, Walker UA, Chung L, Collier DH, Ellen Csuka M, Fessler BJ, Guiducci S, Herrick A, Hsu VM, Jimenez S, Kahaleh B, Merkel PA, Sierakowski S, Silver RM, Simms RW, Varga J, Pope JE. 2013 classification criteria for systemic sclerosis: an American college of rheumatology/European league against rheumatism collaborative initiative. Ann Rheum Dis. 2013 Nov;72(11):1747-55. doi: 10.1136/annrheumdis-2013-204424. PMID 24092682
- [Result] Steele R, Hudson M, Lo E, Baron M; Canadian Scleroderma Research Group. Clinical decision rule to predict the presence of interstitial lung disease in systemic sclerosis. Arthritis Care Res (Hoboken). 2012 Apr;64(4):519-24. doi: 10.1002/acr.21583. PMID 22213733
- [Result] Nihtyanova SI, Schreiber BE, Ong VH, Rosenberg D, Moinzadeh P, Coghlan JG, Wells AU, Denton CP. Prediction of pulmonary complications and long-term survival in systemic sclerosis. Arthritis Rheumatol. 2014 Jun;66(6):1625-35. doi: 10.1002/art.38390. PMID 24591477
- [Result] Denton CP, Khanna D. Systemic sclerosis. Lancet. 2017 Oct 7;390(10103):1685-1699. doi: 10.1016/S0140-6736(17)30933-9. Epub 2017 Apr 13. PMID 28413064
- [Result] Suliman YA, Dobrota R, Huscher D, Nguyen-Kim TD, Maurer B, Jordan S, Speich R, Frauenfelder T, Distler O. Brief Report: Pulmonary Function Tests: High Rate of False-Negative Results in the Early Detection and Screening of Scleroderma-Related Interstitial Lung Disease. Arthritis Rheumatol. 2015 Dec;67(12):3256-61. doi: 10.1002/art.39405. PMID 26316389
- [Result] Tyndall AJ, Bannert B, Vonk M, Airo P, Cozzi F, Carreira PE, Bancel DF, Allanore Y, Muller-Ladner U, Distler O, Iannone F, Pellerito R, Pileckyte M, Miniati I, Ananieva L, Gurman AB, Damjanov N, Mueller A, Valentini G, Riemekasten G, Tikly M, Hummers L, Henriques MJ, Caramaschi P, Scheja A, Rozman B, Ton E, Kumanovics G, Coleiro B, Feierl E, Szucs G, Von Muhlen CA, Riccieri V, Novak S, Chizzolini C, Kotulska A, Denton C, Coelho PC, Kotter I, Simsek I, de la Pena Lefebvre PG, Hachulla E, Seibold JR, Rednic S, Stork J, Morovic-Vergles J, Walker UA. Causes and risk factors for death in systemic sclerosis: a study from the EULAR Scleroderma Trials and Research (EUSTAR) database. Ann Rheum Dis. 2010 Oct;69(10):1809-15. doi: 10.1136/ard.2009.114264. Epub 2010 Jun 15. PMID 20551155
- [Result] Kowal-Bielecka O, Fransen J, Avouac J, Becker M, Kulak A, Allanore Y, Distler O, Clements P, Cutolo M, Czirjak L, Damjanov N, Del Galdo F, Denton CP, Distler JHW, Foeldvari I, Figelstone K, Frerix M, Furst DE, Guiducci S, Hunzelmann N, Khanna D, Matucci-Cerinic M, Herrick AL, van den Hoogen F, van Laar JM, Riemekasten G, Silver R, Smith V, Sulli A, Tarner I, Tyndall A, Welling J, Wigley F, Valentini G, Walker UA, Zulian F, Muller-Ladner U; EUSTAR Coauthors. Update of EULAR recommendations for the treatment of systemic sclerosis. Ann Rheum Dis. 2017 Aug;76(8):1327-1339. doi: 10.1136/annrheumdis-2016-209909. Epub 2016 Nov 9. PMID 27941129
- [Result] Willems LM, Vriezekolk JE, Schouffoer AA, Poole JL, Stamm TA, Bostrom C, Kwakkenbos L, Vliet Vlieland TP, van den Ende CH. Effectiveness of Nonpharmacologic Interventions in Systemic Sclerosis: A Systematic Review. Arthritis Care Res (Hoboken). 2015 Oct;67(10):1426-39. doi: 10.1002/acr.22595. PMID 25832447
- [Result] Avouac J, Walker U, Tyndall A, Kahan A, Matucci-Cerinic M, Allanore Y; EUSTAR; Miniati I, Muller A, Iannone F, Distler O, Becvar R, Sierakowsky S, Kowal-Bielecka O, Coelho P, Cabane J, Cutolo M, Shoenfeld Y, Valentini G, Rovensky J, Riemekasten G, Vlachoyiannopoulos P, Caporali R, Jiri S, Inanc M, Zimmermann Gorska I, Carreira P, Novak S, Czirjak L, Oliveira Ramos F, Jendro M, Chizzolini C, Kucharz EJ, Richter J, Cozzi F, Rozman B, Mallia CM, Gabrielli A, Farge D, Kiener HP, Schoffel D, Airo P, Wollheim F, Martinovic D, Trotta F, Jablonska S, Reich K, Bombardieri S, Siakka P, Pellerito R, Bambara LM, Morovic-Vergles J, Denton C, Hinrichs R, Van den Hoogen F, Damjanov N, Kotter I, Ortiz V, Heitmann S, Krasowska D, Seidel M, Hasler P, Van Laar JM, Kaltwasser JP, Foeldvari I, Juan Mas A, Bajocchi G, Wislowska M, Pereira Da Silva JA, Jacobsen S, Worm M, Graniger W, Kuhn A, Stankovic A, Cossutta R, Majdan M, Damjanovska Rajcevska L, Tikly M, Nasonov EL, Steinbrink K, Herrick A, Muller-Ladner U, Dinc A, Scorza R, Sondergaard K, Indiveri F, Nielsen H, Szekanecz Z, Silver RM, Antivalle M, Espinosa IB, Garcia de la Pena Lefebvre P, Midtvedt O, Launay D, Valesini F, Tuvik P, Ionescu RM, Del Papa N, Pinto S, Wigley F, Mihai C, Sinziana Capranu M, Sunderkotter C, Jun JB, Alhasani S, Distler JH, Ton E, Soukup T, Seibold J, Zeni S, Nash P, Mouthon L, De Keyser F, Duruoz MT, Cantatore FP, Strauss G, von Mulhen CA, Pozzi MR, Eyerich K, Szechinski J, Keiserman M, Houssiau FA, Roman-Ivorra JA, Krummel-Lorenz B, Aringer M, Westhovens R, Bellisai F, Mayer M, Stoeckl F, Uprus M, Volpe A, Buslau M, Yavuz S, Granel B, Valderilio Feijo A, Del Galdo F, Popa S, Zenone T, Ricardo Machado X, Pileckyte M, Stebbings S, Mathieu A, Tulli A, Tourinho T, Souza R, Acayaba de Toledo R, Stamp L, Solanki K, Veale D, Francisco Marques Neto J, Bagnato GF, Loyo E, Toloza S, Li M, Ahmed Abdel Atty Mohamed W, Cobankara V, Olas J, Salsano F, Oksel F, Tanaseanu CM, Foti R, Ancuta C, Vonk M, Caramashi P, Beretta L, Balbir A, Chiala A, Pasalic Simic K, Ghio M, Stamenkovic B, Rednic S, Host N, Pellerito R, Hachulla E, Furst DE. Characteristics of joint involvement and relationships with systemic inflammation in systemic sclerosis: results from the EULAR Scleroderma Trial and Research Group (EUSTAR) database. J Rheumatol. 2010 Jul;37(7):1488-501. doi: 10.3899/jrheum.091165. Epub 2010 Jun 15. PMID 20551097
- [Result] Clements PJ, Furst DE, Campion DS, Bohan A, Harris R, Levy J, Paulus HE. Muscle disease in progressive systemic sclerosis: diagnostic and therapeutic considerations. Arthritis Rheum. 1978 Jan-Feb;21(1):62-71. doi: 10.1002/art.1780210111. PMID 623695
- [Result] Lima TR, Guimaraes FS, Carvalho MN, Sousa TL, Menezes SL, Lopes AJ. Lower limb muscle strength is associated with functional performance and quality of life in patients with systemic sclerosis. Braz J Phys Ther. 2015 Mar-Apr;19(2):129-36. doi: 10.1590/bjpt-rbf.2014.0084. Epub 2015 Mar 13. PMID 25789555
- [Result] Blom-Bulow B, Jonson B, Bauer K. Factors limiting exercise performance in progressive systemic sclerosis. Semin Arthritis Rheum. 1983 Nov;13(2):174-81. doi: 10.1016/0049-0172(83)90004-5. PMID 6673113
- [Result] Cuomo G, Santoriello C, Polverino F, Ruocco L, Valentini G, Polverino M. Impaired exercise performance in systemic sclerosis and its clinical correlations. Scand J Rheumatol. 2010 Aug;39(4):330-5. doi: 10.3109/03009740903555358. PMID 20476863
- [Result] de Oliveira NC, dos Santos Sabbag LM, Ueno LM, de Souza RB, Borges CL, de Sa Pinto AL, Lima FR. Reduced exercise capacity in systemic sclerosis patients without pulmonary involvement. Scand J Rheumatol. 2007 Nov-Dec;36(6):458-61. doi: 10.1080/03009740701605889. PMID 18092268
- [Result] Hudson M, Thombs BD, Steele R, Panopalis P, Newton E, Baron M; Canadian Scleroderma Research Group. Health-related quality of life in systemic sclerosis: a systematic review. Arthritis Rheum. 2009 Aug 15;61(8):1112-20. doi: 10.1002/art.24676. PMID 19644906
- [Result] Oliveira NC, dos Santos Sabbag LM, de Sa Pinto AL, Borges CL, Lima FR. Aerobic exercise is safe and effective in systemic sclerosis. Int J Sports Med. 2009 Oct;30(10):728-32. doi: 10.1055/s-0029-1224180. Epub 2009 Jul 29. PMID 19642060
- [Result] Holland AE. Exercise limitation in interstitial lung disease - mechanisms, significance and therapeutic options. Chron Respir Dis. 2010;7(2):101-11. doi: 10.1177/1479972309354689. Epub 2010 Jan 7. PMID 20056733
- [Result] Holland A, Hill C. Physical training for interstitial lung disease. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD006322. doi: 10.1002/14651858.CD006322.pub2. PMID 18843713
- [Result] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Result] Graham BL, Brusasco V, Burgos F, Cooper BG, Jensen R, Kendrick A, MacIntyre NR, Thompson BR, Wanger J. 2017 ERS/ATS standards for single-breath carbon monoxide uptake in the lung. Eur Respir J. 2017 Jan 3;49(1):1600016. doi: 10.1183/13993003.00016-2016. Print 2017 Jan. PMID 28049168
- [Result] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257